CLINICAL TRIAL: NCT06452667
Title: Platelet Rich Fibrin Versus Platelet Rich Plasma for Microneedling Treatment of Facial Photoaging-a Double Blind Randomized Controlled Study
Brief Title: Platelet Rich Fibrin Versus Platelet Rich Plasma for Microneedling Treatment of Facial Photoaging
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yau-Li Huang, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPRPG5P0011
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Photoaging
Keywords: photoaging; platelet rich plasma; Platelet rich fibrin

STUDY DESIGN:
Intervention Model Description: Each case will receive 3 sessions of injection therapies with one month interval (T0, T1, and T2). Each case will receive PRP therapy on one side of the face. The other side of the face was treated with platelet-rich fibin (PRF).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization numbers will be generated via SAS software version 9.4 by independent blinded personnel outside our research team. We will use the randomization numbers to determine the treatment method for both sides of each case before the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet-rich fibin (Experimental): Each case will receive 3 sessions of therapies with one month interval. We will apply 1-2ml PRF to the photoaging areas in one side of the cheek of patients by using microneedling.
  Interventions: Procedure: platelet-rich fibin
- platelet-rich palsma (Active Comparator): Each case will receive 3 sessions of therapies with one month interval. We will apply 1-2ml PRP to the photoaging areas in one side of the cheek of patients by using microneedling.
  Interventions: Procedure: platelet-rich palsma

INTERVENTIONS:
Procedure: platelet-rich fibin — Each case will receive 3 sessions of microneedling therapies with one month interval. Each case will receive platelet-rich fibin therapy on one side of the face. The other side of the face was treated with platelet-rich palsma.
  Arms: platelet-rich fibin
Procedure: platelet-rich palsma — Each case will receive 3 sessions of microneedling therapies with one month interval. Each case will receive platelet-rich palsma therapy on one side of the face. The other side of the face was treated with platelet-rich fibin.
  Arms: platelet-rich palsma

SUMMARY:
The present study was conducted for analyzing the efficacy and safety of platelet-rich plasma (PRP) and platelet-rich fibrin (PRF) in photoaging therapy.

Specific arms:

1. The investigators will compare the photoaging improvement of PRF and PRP treated face before and after treatment by two blinded investigators.
2. The investigators will evaluate the improvement of each parameter of photoaging by Visia system, dermoscope, and optical coherence tomography.
3. The investigators will evaluate the safety of the treatment of PRF and PRP.

Each case will receive 3 sessions of injection therapies with one month interval (T0, T1, and T2). Each case will receive PRP therapy on one side of the face and PRF on the other side of face. The investigators will determine the treatment method for both sides of each case randomly by coin flapping before the study. The investigators will evaluate each case before each session of therapy (T0, T1, T2) as well as 1 (T3) and 3 months (T4) after final session of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men or female patients older than 20 years old with facial photoaging (Glogau Scale type II)
2. The photoaging severity of bilateral face is symmetric.

Exclusion Criteria:

1. Patients with thrombocytopenia, coagulopathy, hematopoietic malignancy.
2. Patients with severe inflammation over treated area, malignancy, keloid, or poor wound healing history.
3. Patients had received laser, radiofrequency, ultherapy over treated area within 6 months.
4. Patients had received botulism or filler injection over treated area within 12 months.
5. Patients had received plastic surgery over treated area within 12 months.
6. Patients had severe psychiatric disorders with poor control.
7. Patients with other diseases which are not suitable for receiving platelet rich plasma (PRP) or platelet rich fibrin (PRF) therapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Global Aesthetic Improvement Scale | 3 months after the last session of treatment
  We will compare the photoaging improvement of PRF and PRP treated face before treatment and 3 months after last treatment by two blinded investigators using Global Aesthetic Improvement Scale (GAIS). GAIS, which is a 5-point scale wherein 5 = very much improved, 4 = much improved, 3 = improved, 2 = no change, and 1= worse.

SECONDARY OUTCOMES:
Fitzpatrick wrinkle scale | 3 months after the last session of treatment
  To assess the severity of wrinkles of photoaging areas (minimum: 1, mild; maximum: 9, severe)
Wrinkle Severity Rating scale | 3 months after the last session of treatment
  To assess the severity of wrinkles of photoaging areas (minimum: 1, absent; maximum: 5, extreme)

OTHER OUTCOMES:
The scores of rhytids in VISIA system | 3 months after the last session of treatment
  Apply the scores of different aging domains in VISIA system for evaluating the therapeutic response. (minimum: 1, worse; maximum: 100, severe)
The scores of Textures in VISIA system | 3 months after the last session of treatment
  Apply the scores of different aging domains in VISIA system for evaluating the therapeutic response. (minimum: 1, worse; maximum: 100, severe)
The scores of Pores size in VISIA system | 3 months after the last session of treatment
  Apply the scores of different aging domains in VISIA system for evaluating the therapeutic response. (minimum: 1, worse; maximum: 100, severe)
The scores of Brown spots in VISIA system | 3 months after the last session of treatment
  Apply the scores of different aging domains in VISIA system for evaluating the therapeutic response. (minimum: 1, worse; maximum: 100, severe)
The scores of Spots in VISIA system | 3 months after the last session of treatment
  Apply the scores of different aging domains in VISIA system for evaluating the therapeutic response. (minimum: 1, worse; maximum: 100, severe)
The scores of UV spots in VISIA system | 3 months after the last session of treatment
  Apply the scores of different aging domains in VISIA system for evaluating the therapeutic response. (minimum: 1, worse; maximum: 100, severe)
The scores of red areas in VISIA system | 3 months after the last session of treatment
  Apply the scores of different aging domains in VISIA system for evaluating the therapeutic response. (minimum: 1, worse; maximum: 100, severe)
Dermoscopy Photoaging Scale | 3 months after the last session of treatment
  Photoaging evaluation instrument using a dermoscopy (minimum: 0, worse; maximum: 11, severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
We will not share IPD due to the privacy of participants.

REFERENCES:
- [Result] Lee ZH, Sinno S, Poudrier G, Motosko CC, Chiodo M, Saia W, Gothard D, Thomson JE, Hazen A. Platelet rich plasma for photodamaged skin: A pilot study. J Cosmet Dermatol. 2019 Feb;18(1):77-83. doi: 10.1111/jocd.12676. Epub 2018 May 31. PMID 29855132
- [Result] Mahmoodabadi RA, Golafshan HA, Pezeshkian F, Shahriarirad R, Namazi MR. Evaluation of the Effect of Platelet-Rich Fibrin Matrix in the Correction of Periorbital Wrinkles: An Experimental Clinical Trial. Dermatol Pract Concept. 2023 Jan 1;13(1):e2023050. doi: 10.5826/dpc.1301a50. PMID 36892335
- [Result] Hassan H, Quinlan DJ, Ghanem A. Injectable platelet-rich fibrin for facial rejuvenation: A prospective, single-center study. J Cosmet Dermatol. 2020 Dec;19(12):3213-3221. doi: 10.1111/jocd.13692. Epub 2020 Sep 23. PMID 32852873
- [Result] Isik B, Gurel MS, Erdemir AT, Kesmezacar O. Development of skin aging scale by using dermoscopy. Skin Res Technol. 2013 May;19(2):69-74. doi: 10.1111/srt.12033. Epub 2013 Jan 20. PMID 23331299
- [Result] Evans AG, Ivanic MG, Botros MA, Pope RW, Halle BR, Glassman GE, Genova R, Al Kassis S. Rejuvenating the periorbital area using platelet-rich plasma: a systematic review and meta-analysis. Arch Dermatol Res. 2021 Nov;313(9):711-727. doi: 10.1007/s00403-020-02173-z. Epub 2021 Jan 12. PMID 33433716
- [Result] Salminen A, Kaarniranta K, Kauppinen A. Photoaging: UV radiation-induced inflammation and immunosuppression accelerate the aging process in the skin. Inflamm Res. 2022 Aug;71(7-8):817-831. doi: 10.1007/s00011-022-01598-8. Epub 2022 Jun 24. PMID 35748903
- [Result] Diab NAF, Ibrahim AM, Abdallah AM. Fluid Platelet-Rich Fibrin (PRF) Versus Platelet-Rich Plasma (PRP) in the Treatment of Atrophic Acne Scars: A Comparative Study. Arch Dermatol Res. 2023 Jul;315(5):1249-1255. doi: 10.1007/s00403-022-02511-3. Epub 2022 Dec 15. PMID 36520210